CLINICAL TRIAL: NCT01494987
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Ranolazine When Added to Glimepiride in Subjects With Type 2 Diabetes Mellitus
Brief Title: Ranolazine When Added to Glimepiride in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-259-0110
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ranolazine; glimepiride; Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine+glimepiride (Experimental): Glimepiride stabilization period (up to 8 weeks): participants not on stable glimepiride will receive glimepiride 2 mg once daily, and if tolerated the dose will be increased on Day 8 (+ 2 days) to 4 mg once daily.
  Qualifying period: participants will receive placebo to match ranolazine twice daily in addition to glimepiride for 14 days (+ 2 days) and if ≥ 80% compliant and meeting eligibility criteria will continue to the treatment period.
  Treatment period: participants will be randomized to receive ranolazine 500 mg twice daily plus glimepiride 4 mg once daily on Days 1 through 7, followed by ranolazine 1000 mg twice daily plus glimepiride 4 mg once daily from Day 8 (or by Day 16 if not well tolerated) through Week 24.
  Participants will be required to maintain their diet and exercise regimen.
  Interventions: Drug: Ranolazine; Drug: Glimepiride; Behavioral: Diet; Behavioral: Exercise
- Placebo+glimepiride (Placebo Comparator): Glimepiride stabilization period (up to 8 weeks): participants not on stable glimepiride will receive glimepiride 2 mg once daily, and if tolerated the dose will be increased on Day 8 (+ 2 days) to 4 mg once daily.
  Qualifying period: participants will receive placebo to match ranolazine twice daily in addition to glimepiride for 14 days (+ 2 days) and if ≥ 80% compliant and meeting eligibility criteria will continue to the treatment period.
  Treatment period: participants will be randomized to receive placebo to match ranolazine plus glimepiride 4 mg once daily for 24 weeks.
  Participants will be required to maintain their diet and exercise regimen.
  Interventions: Drug: Placebo; Drug: Glimepiride; Behavioral: Diet; Behavioral: Exercise

INTERVENTIONS:
Drug: Ranolazine — Ranolazine tablet(s) administered orally
  Other Names: Ranexa®
  Arms: Ranolazine+glimepiride
Drug: Placebo — Placebo to match ranolazine for the duration of the study
  Arms: Placebo+glimepiride
Drug: Glimepiride — Glimepiride tablets (2 mg or 4 mg) administered orally once daily with the morning dose of study drug or placebo. The target dosing regimen for glimepiride is 4 mg once daily.
Behavioral: Diet — Participants are instructed to continue the diet regimen prescribed by their physician.
Behavioral: Exercise — Participants are instructed to continue the exercise regimen prescribed by their physician.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, multi-center study to determine the effect of ranolazine when added to glimepiride on glycemic control in adults with type 2 diabetes mellitus (T2DM) who are inadequately controlled despite current treatment with stable sulfonylurea or metformin therapy in addition to diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Males and females, 18 to 75 years old, inclusive
* Documented history of T2DM
* Receiving one of the following sulfonylurea or metformin therapies in addition to diet and exercise for at least 90 days prior to Screening:

  1. glimepiride at a daily dose of ≥ 2 mg and ≤ 4 mg
  2. glipizide, glyburide, or glibenclamide (or equivalent) at a daily dose of ≥ 7.5 mg
  3. gliclazide at a daily dose of > 160 mg (or ≥ 60 mg for the modified release [MR] formulation)
  4. metformin at a daily dose of ≥ 1500 mg
* Body mass index (BMI) 25 kg/m2 to 45 kg/m2, inclusive, at Screening
* HbA1c 7% to 10%, inclusive, at Screening and the end of the Qualifying Period (Day 14)
* Fasting Serum C-peptide ≥ 0.8 ng/mL at Screening
* Fasting serum glucose (FSG) ≥ 130 mg/dL (7.2 mmol/L) and ≤ 240 mg/dL (13.3 mmol/L) at Screening and at the end of the Qualifying Period (Day 14): A one-time central laboratory re-test of FSG is allowed in subjects with an initial central laboratory FSG ≥ 120 mg/dL (6.7 mmol/L) and < 130 mg/dL (7.2 mmol/L) who are otherwise eligible as determined by the investigator.
* Able and willing to comply with all study procedures during the course of the study
* Females of child-bearing potential must have a negative serum pregnancy test at Screening and must agree to use highly effective contraception methods from Screening throughout the duration of the Treatment Period and for 14 days following the last dose of study drug.
* At least 80% compliant in dosing during the Qualifying Period

Exclusion Criteria:

* History of or current diagnosis of type 1 diabetes mellitus
* History of diabetic ketoacidosis, ketosis-prone diabetes, or hyperosmolar hyperglycemic coma
* History of a severe episode of hypoglycemia (≥ 1 episode within 3 months prior to Screening or ≥ 2 episodes within 6 months prior to Screening), defined as hypoglycemia requiring 3rd party assistance to actively administer carbohydrate, glucagon, or other resuscitative actions due to severe impairment in consciousness or behavior
* Clinically significant complications of diabetes that in the judgment of the investigator would make the subject unsuitable to participate in this study
* History of any clinically significant cardiovascular (CV) or cerebrovascular event (eg, myocardial infarction [MI], acute coronary syndrome [ACS], recent revascularization [including coronary artery bypass graft procedures or percutaneous coronary intervention], transient ischemic attack, or ischemic stroke) ≤ 3 months prior to Screening
* Inadequately controlled or unstable hypertension as defined by a systolic blood pressure (SBP) > 160 mmHg or diastolic blood pressure (DBP) > 100 mmHg at Screening and at Randomization
* Prolonged QT interval corrected for heart rate (QTc) interval > 500 msec by electrocardiogram (ECG) at Screening, a personal or family history of QTc prolongation, congenital long QT syndrome, or subjects who are receiving drugs that prolong the QTc interval, such as Class Ia or Class III antiarrhythmic agents, erythromycin, and certain antipsychotics (eg, ziprasidone)
* History of bariatric surgery at any time in the past or or any other surgery < 2 months before Screening; or planning to undergo surgery during the study. Subjects with a planned minor surgery may be enrolled upon approval by the medical monitor.
* Any other hospitalization in the 14 days prior to Screening or planned hospitalization at any time during the study
* Significant weight change (± 5%) < 2 months prior to Screening or enrollment in a weight-loss program other than a maintenance phase at Screening.
* Severe renal impairment, defined as an estimated glomerular filtration rate (eGFR) by the Modification of Diet in Renal Disease (MDRD) equation < 30 mL/min/1.73 m2 at Screening or undergoing any type of dialysis at Screening or planning to undergo any type of dialysis during the course of the study
* History of liver cirrhosis (Child-Pugh Class A, B or C)
* Active liver disease and/or significant abnormal liver function defined as aspartate aminotransferase (AST) > 3 x upper limit of the normal range (ULN) and/or alanine aminotransferase (ALT) > 3 x ULN and/or serum total bilirubin > 2.0 mg/dL
* History of cancer (except nonmelanomic skin cancers or cervical in situ) within 5 years prior to Screening
* History of alcohol or other drug abuse < 12 months prior to Screening
* Any other clinically significant existing medical or psychiatric condition, including clinically significant laboratory abnormalities, or one requiring further evaluation that in the opinion of the investigator could interfere with conduct of the study or interpretation of the data
* Use of antihyperglycemic agents other than sulfonylurea agents or metformin, including but not limited to dipeptidyl peptidase-4 inhibitors (eg, saxagliptin and sitagliptin), glucagon-like peptide-mimetics (eg, exenatide), or insulin < 3 months prior to Screening; use of thiazolidinediones (TZDs) (eg, rosiglitazone or pioglitazone) < 24 weeks prior to Screening
* Previous history of intolerance of glimepiride (as a single-agent therapy)
* Prior treatment with open-label ranolazine, or known hypersensitivity or intolerance to ranolazine or any of its excipients
* Treatment with strong or moderate cytochrome P (CYP)3A inhibitors or P-glycoprotein (P-gp) inhibitors within 14 days prior to randomization
* Treatment with CYP3A inducers or P-gp inducers within 14 days prior to randomization
* Treatment with CYP3A4 substrates with a narrow therapeutic range (eg, cyclosporine, tacrolimus, or sirolimus) within 14 days prior to Randomization
* Treatment with simvastatin at a dose of > 20 mg daily or lovastatin at a dose of > 40 mg daily within 14 days prior to Randomization
* Weight loss medication or anti-obesity medication (prescription or non-prescription) < 3 months prior to Screening
* Treatment with niacin > 200 mg daily; if receiving ≤ 200 mg daily, should be on stable doses for ≥ 3 months prior to Screening
* Expected or current treatment with systemic corticosteroids (oral or injectable) for > 14 days from Screening through the end of the Treatment Period. Topical or inhaled corticosteroid formulations are permitted at any time during the study.
* If receiving thyroid replacement therapy, should be on stable doses for at least 6 weeks prior to randomization
* Hemoglobin < 12 g/dL for males or < 11 g/dL for females at Screening
* Participation in another clinical study involving an investigational drug or device < 30 days prior to Screening; participation in another clinical study involving an oral antihyperglycemic agent (OHA) < 90 days prior to Screening
* Donation of blood < 2 months prior to Screening or plans to donate blood while participating in the study
* Females who are pregnant or are breastfeeding
* Other condition(s) that, in the opinion of the investigator, would compromise the safety of the individual, prevent compliance with the study protocol (including the ability to comply with Mixed Meal Tolerance Test [MMTT]), or compromise the quality of the clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yue, MD, Study Director — Gilead Sciences
Locations (139):
- United States (45):
  - Clinical Research Advantage/Desert Clinical Research, LLC, Mesa, Arizona
  - Desert Sun Clinical Research, LLC, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Paul W. Davis, MD, PA, Pine Bluff, Arkansas
  - Southland Clinical Research Center, Inc., Fountain Valley, California
  - Valley Research, Fresno, California
  - Del Rosario Medical Clinic, Inc., Huntington Park, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - National Research Institute, Los Angeles, California
  - Spectrum Clinical Research Institute, Inc, Moreno Valley, California
  - Sacramento Heart and Vascular Medical Associates, Sacramento, California
  - Infosphere Clinical Research, West Hills, California
  - PAB Clinical Research, Brandon, Florida
  - Florida Research Network, LLC, Gainesville, Florida
  - NewPhase Clinical Trials, Inc., Miami Beach, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Regenerate Clinical Trials, South Miami, Florida
  - Comprehensive Clinical Development, Inc., St. Petersburg, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Synergy Therapeutic Partners, Atlanta, Georgia
  - CTL Research, Eagle, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - LaPorte County Institute for Clinical Research, Michigan City, Indiana
  - L-MARC Research Center, Louisville, Kentucky
  - Horizon Research Group of Opelousas, Eunice, Louisiana
  - MD Medical Research, Oxon Hill, Maryland
  - IRC Clinics, Inc, Towson, Maryland
  - Endeavor Medical Research, PLC, Alpena, Michigan
  - Associated Internal Medicine Specialists, P.C., Battle Creek, Michigan
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - PMG Research of Charlotte, Charlotte, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Clinical Inquest Center, Ltd., Beavercreek, Ohio
  - Infinity Research Group, LLC, Oklahoma City, Oklahoma
  - Southeastern Research Associates, Inc., Taylors, South Carolina
  - HCCA Clinical Research Solution, Franklin, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Excel Clinical Research, LLC, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Humble Cardiology Associates, Humble, Texas
  - Cetero Research, San Antonio, Texas
  - Highland Clinical Research, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah
- Interni oddeleni, Havířov, Moravskoslezský kraj, Czechia
- Hungary (6):
  - Drug Research Center, Balatonfüred
  - Synexus Hungary Ltd, Budapest
  - Markhot Ferenc Hospital, Eger
  - Kanizsai Dorottya Hospital, Nagykanizsa
  - Borbanya Praxis Kft., Outpatient Clinic, Nyíregyháza
  - Medifarma 98, Nyíregyháza
- Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia
- Poland (8):
  - NZOZ Centrum Badan Klinicznych, Wroclaw, Lower Silesian Voivodeship
  - Centrum Badan Klinicznych PI-House Sp. z o.o., Gdansk, Pomeranian Voivodeship
  - LANDA - Specjalistyczne Gabinety Lekarskie, Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny Nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Łodzi, Oddział Kliniczny Diabetologii, Lodz
  - NZOZ Centrum Badan Klinicznych Oswiecim, Oswięcim
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska Sp. Komandytowo - Akcyjna, Lodz, Łódź Voivodeship
  - NZOZ Centrum Medyczne Szpital Sw. Rodziny, Lodz, Łódź Voivodeship
  - NZOZ Polimedica, Zgierz, Łódź Voivodeship
- Romania (11):
  - CMI Morosanu V. Magdalena, Galati, Galați County
  - Spital Clinic Judetean de Urgenta Oradea Stationarul 1, Oradea, Jud Bihor
  - Consultmed SRL, Iași, Jud. Iasi
  - Centru Medical Dr. Negrisanu, Timișoara, Judical Timis
  - Institutul de Diabet, Nutritie si Boli Metabolice "Dr. N. C. Paulescu", Bucharest
  - Tehnomed Trading Srl, Bucharest
  - Institutul National De Diabet, Nutritie Si Boli Metabolice "Prof. Dr. N.C. Paulescu", Bucharest
  - O.D. Medica Srl, Bucharest
  - CMI Mateescu S. Ana-Maria, Constanța
  - Spitalul Clinic Judetean de Urgenta "Sf. Apostol Andrei" Galati, Galati
  - Diabmed Dr. Popescu Alexandrina SRL, Ploieşti
- Russia (36):
  - 3rd Central Military Clinical Hospital named after A.A.Vishnevskogo, Arkhangel'skoye
  - GOU VPO "Chita State Medical Academy" of Minzdravsocrazvitie RF, Chita
  - "Clinic of New Medical Technology" Company Limited, Dzerzhinskiy
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - "Krasnoyarsk State Medical University n.a. Prof. V.F. Voyno-Yasenetsky, Krasnoyarsk
  - State Healthcare Institution of Moscow "Cardiologival Dispensary #2 of Management Department of South Administrative District", Moscow
  - Central Clinical Hospital of Russian Academy of Sciences, Moscow
  - Medical Sanitary Unit of Minestry of Internal Affairs of Russia in Moscow, Moscow
  - City Clinical Hospital # 13 of Avtozavodsky District of Nizhniy Novgorod, Nizhny Novgorod
  - Novosibirsk State Medical University, Novosibirsk
  - Scientific Research Institute of Physiology of Siberian Department RAMS, Novosibirsk
  - City Hospital # 38 named after N A Semashko, Pushkin
  - Rostov State Medical University, Rostov-on-Don
  - Ryazan State Medical University, Ryazan
  - Medinet, LLC, Saint Petersburg
  - North-Western State Medical Unversity n.a. I.I.Mechnikov, Saint Petersburg
  - Saint-Petersburg City Outpatient Clinic#37, Saint Petersburg
  - Military Medical Academy named after S.M. Kirov, Saint Petersburg
  - Saint-Petersburg state budgetary healthcare institution "City Polyclinic #109", Saint Petersburg
  - Alexanders City Hospital, Saint Petersburg
  - Clinical Hospital #122 n.a. Sokolov of FMBA, Saint Petersburg
  - ANO "Medical Centre "XXI century", Saint Petersburg
  - St. Elizabeth City Hospital, Saint Petersburg
  - Krestovsky Island Medical Institute, LLC, Saint Petersburg
  - Federal Centre of Heart, Blood and Endocrinology named after V.A. Almazov, Saint Petersburg
  - International Medical Center "SOGAZ", LLC, Saint Petersburg
  - Saint-Petersburg City Pokrovskaya Hospital, Saint Petersburg
  - Center "Diabetes", LLC, Samara
  - Smolensk State Medical Academy, Sanatorium-Preventorium, Smolensk
  - Tyumen State Medical Academy, Tyumen
  - Voronezh Regional Clinical Hospital #1, Voronezh
  - City Hospital named after N.A.Semashko, Yaroslavl
  - Clinical Hospital for Emergency Care named after N.V. Solovyov, Yaroslavl
  - Medical Sanitary Unit of Novo-Yaroslavsky Oil Refinery, Yaroslavl
  - Yaroslavl Regional Clinical Hospital, Yaroslavl
  - The Urals State Medical Academy, Yekaterinburg
- Serbia (3):
  - Clinical Center of Serbia, Belgrade
  - Zvezdara University Medical Center, Belgrade
  - Clinical Center of Kragujevac, Kragujevac
- Slovakia (5):
  - METABOLKLINIK s.r.o., Bratislava, Bratislava Region
  - Metabolic Center of Dr. Katarina Raslova Ltd., Bratislava, Bratislava Region
  - ARETEUS s.r.o., Diabetologicka ambulancia, Trebišov, Košice Region
  - MediVet s.r.o., Malacky
  - ENDIAMED s.r.o, Dolný Kubín, Žilina Region
- South Africa (10):
  - Newkwa Medical Centre, Newlands West, Durban
  - Drs. Naiker and Naicker Inc., Overport, Durban
  - Centre for Diabetes and Endocrinology Suite 1, Durban
  - Centre for Diabetes, Asthma and Allergy, Johannesburg
  - Soweto Clinical Trial Centre, Johannesburg
  - Centre fro Diabetes and Endocrinology (Pty) Ltd, Johannesburg
  - Aliwal Shoal Medical & Clinical Trial Centre, Kwa Zulu Natal
  - Paarl Research Centre, Paarl, Cape Town
  - Helderberg Clinical Trials Centre, Somerset West
  - Tiervlei Trial Centre, Western Cape
- Thailand (4):
  - Chulalongkorn University, Patumwan, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Songklanagarind Hospital, Songkhla
- Ukraine (9):
  - City Clinical Hospital#9, Dnipropetrovsk State Medical Academy, Dnipropetrovsk
  - Educational Scientific Medical Centre "University clinic" of Donetsk National Medical University n.a. M.Gorkiy, Donetsk
  - Administration of Medical Service and Rehabilitation of "ARTEM" State Holding Company, Kyiv
  - National Medical University n.a. O.O. Bogomolets, Chair of Family Medicine based on Outpatient Clinic # 2 of Shevchenkovsky District, Kyiv
  - V. P. Komissarenko Institute of Endocrinology and Metabolism of AMS of Ukraine, Kyiv
  - Municipal Institution Lutsk City Clinical Hospital, Lutsk
  - Lviv Regional Endocrinology Dispensary, Lviv
  - Odessa State Medical University, Odesa
  - Zhytomyr Regional Clinical Hospital, Zhytomyr

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled (during the Qualifying Period) at a total of 103 study sites in Asia, Europe, South Africa, and the United States. The first participant was screened on 12 January 2012. The last participant observation occurred on 28 August 2013.
Pre-assignment Details: 595 participants entered the qualifying period (355 required and completed the glimepiride stabilization period); 431 were randomized and treated (Safety Analysis Set). Of these, 14 were excluded due to major eligibility criteria protocol violation or had no baseline or ontreatment data; thus, 417 were included in the Full Analysis Set.
Groups:
- Placebo+Glimepiride: Glimepiride stabilization period (up to 8 weeks): participants not on stable glimepiride received glimepiride 2 mg once daily, and if tolerated the dose was increased on Day 8 (+ 2 days) to 4 mg once daily.
  Qualifying period: participants received placebo to match ranolazine twice daily in addition to glimepiride for 14 days (+ 2 days) and if ≥ 80% compliant and meeting eligibility criteria continued to the treatment period.
  Treatment period: participants were randomized to receive placebo to match ranolazine plus glimepiride 4 mg once daily for 24 weeks.
  Participants were required to maintain their diet and exercise regimen.
- Ranolazine+Glimepiride: Glimepiride stabilization period (up to 8 weeks): participants not on stable glimepiride received glimepiride 2 mg once daily, and if tolerated the dose was increased on Day 8 (+ 2 days) to 4 mg once daily.
  Qualifying period: participants received placebo to match ranolazine twice daily in addition to glimepiride for 14 days (+ 2 days) and if ≥ 80% compliant and meeting eligibility criteria continued to the treatment period.
  Treatment period: participants were randomized to receive ranolazine (1 x 500 mg tablet) twice daily plus glimepiride 4 mg once daily on Days 1 through 7, followed by ranolazine 1000 mg (2 x 500 mg tablets) twice daily plus glimepiride 4 mg once daily from Day 8 (or by Day 16 if not well tolerated) through Week 24.
  Participants were required to maintain their diet and exercise regimen.
Period: Overall Study
Arm/Group | Placebo+Glimepiride | Ranolazine+Glimepiride
Started | 216 | 215
Completed | 188 | 187
Not Completed | 28 | 28
Not completed — Adverse Event | 6 | 5
Not completed — Hyperglycemia | 6 | 4
Not completed — Investigator's Discretion | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 3 | 3
Not completed — Subject Non-Compliance | 9 | 10
Not completed — Subject Withdrew Consent | 2 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the Safety Analysis Set following randomization. The Safety Analysis Set includes randomized participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo+Glimepiride | Ranolazine+Glimepiride | Total
Number analyzed (Participants) | 216 | 215 | 431
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (8.6) | 59 (8.8) | 59 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 120 | 243
  Male | 93 | 95 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 32 | 64
  Not Hispanic or Latino | 181 | 182 | 363
  Unknown or Not Reported | 3 | 1 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 3 | 7
  Black or African American | 10 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 198 | 204 | 402
  Other | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  Serbia | 4 | 0 | 4
  United States | 61 | 60 | 121
  Czech Republic | 1 | 0 | 1
  Hungary | 4 | 6 | 10
  Slovakia | 1 | 2 | 3
  Poland | 5 | 4 | 9
  Ukraine | 26 | 27 | 53
  Romania | 11 | 9 | 20
  South Africa | 4 | 3 | 7
  Russian Federation | 99 | 104 | 203
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.8 (4.35) | 32.2 (3.88) | 32.5 (4.13)
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent HbA1c in blood] | 8.10 (0.746) | 8.07 (0.776) | 8.08 (0.760)
Fasting Serum Glucose [Mean (Standard Deviation); unit: mg/dL] | 177.2 (34.27) | 177.4 (37.03) | 177.3 (35.63)
Duration of Diabetes [Mean (Standard Deviation); unit: years] — Participants in the Safety Analysis Set with available data were analyzed (n = 215 in both groups).
  years | 7.0 (5.07) | 7.1 (4.92) | 7.0 (4.99)
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 83.2 (18.77) | 81.2 (20.85) | 82.2 (19.84)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: The average (mean) change from baseline in HbA1c at Week 24 was analyzed.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set (randomized participants who received ≥ 1 dose of study treatment with a baseline and at least one postbaseline measurement of HbA1c, excluding participants with major eligibility violations and analyzed based on randomized treatment, regardless of actual treatment received) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent of HbA1c in blood
Arm/Group | Placebo+Glimepiride | Ranolazine+Glimepiride
Number analyzed (Participants) | 184 | 188
percent of HbA1c in blood
  HbA1c at Week 24 | 8.08 (1.070) | 7.58 (1.089)
  Change from baseline in HbA1c at Week 24 | 0.03 (0.949) | -0.47 (0.971)
Statistical Analysis 1: Comparison: Placebo+Glimepiride vs Ranolazine+Glimepiride; Assuming a common standard deviation of 1.2%, an effective sample size of 400 would provide at least 90% power to detect a statistically significant treatment difference of -0.5% (ranolazine vs. placebo) for the reduction of HbA1c from baseline at Week 24 based on a 2-sided alpha of 0.05 and 1:1 randomization; Test type: Superiority or Other; p < 0.001, Mixed Effects Model Analysis — P-value is from a mixed-effect model including terms for baseline HbA1c value, prior antihyperglycemia therapy, treatment group, visit week, and treatment by visit week interaction. Unstructured covariance matrix was used; difference in least squares mean (LSM) = -0.51, 95% CI 2-sided [-0.71 to -0.32] — The estimation (LSM) is of the placebo-corrected change from baseline

2. Secondary Outcome: Change From Baseline in Incremental Change of 2-hour Postprandial Serum Glucose at Week 24
Description: The average (mean) change from baseline in incremental change of 2-hour postprandial serum glucose at Week 24 was analyzed.
  Mixed Meal Tolerance Test (MMTT) Full Analysis Set: randomized participants who received at least one dose of study treatment with a baseline and at least one postbaseline measurement of serum glucose at T=120 minutes during the MMTT, administered under fasting conditions, excluding participants with major eligibility protocol violations, analyzed based on the randomized treatment regardless of actual treatment received.
Time Frame: Baseline; Week 24
Population: Participants in the Mixed Meal Tolerance Test (MMTT) Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo+Glimepiride | Ranolazine+Glimepiride
Number analyzed (Participants) | 169 | 168
mg/dL | -2 (42.6) | 1 (44.7)

3. Secondary Outcome: Change From Baseline in Fasting Serum Glucose at Week 24
Description: The average (mean) change from baseline in fasting serum glucose at Week 24 was analyzed.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo+Glimepiride | Ranolazine+Glimepiride
Number analyzed (Participants) | 181 | 183
mg/dL | 8 (40.7) | 2 (45.3)

4. Secondary Outcome: Change From Baseline in 2-hour Postprandial Serum Glucose at Week 24
Description: The average (mean) change from baseline in 2-hour postprandial serum glucose at Week 24 was analyzed.
Time Frame: Baseline; Week 24
Population: Participants in the MMTT Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo+Glimepiride | Ranolazine+Glimepiride
Number analyzed (Participants) | 175 | 172
mg/dL | 4 (58.0) | 1 (59.6)

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Arm/Group | Placebo+Glimepiride | Ranolazine+Glimepiride
Serious Adverse Events (participants affected / at risk) | 4/216 | 4/215
Other Adverse Events (participants affected / at risk) | 46/216 | 42/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+Glimepiride (N=216) | Ranolazine+Glimepiride (N=215)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 1
Retinal vein thrombosis (Eye disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+Glimepiride (N=216) | Ranolazine+Glimepiride (N=215)
Hyperglycemia (Metabolism and nutrition disorders) | 32 | 21
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 13
Nausea (Gastrointestinal disorders) | 7 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years